CLINICAL TRIAL: NCT05157022
Title: Comparative Effects of Radial and Focused Extracorporeal Shock-wave Therapies in Coccydynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yuzuncu Yıl
Record Dates: First submitted 2021-10-13; First posted 2021-12-14 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Coccyx Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus extracorporeal shock wave therapy (Active Comparator): A total of 4 sessions of ESWT at 1-week intervals were applied to to the sacrococcygeal area
  Interventions: Device: ESWT
- Radial extracorporeal shock wave therapy (Active Comparator): A total of 4 sessions of ESWT at 1-week intervals were applied to to the sacrococcygeal area
  Interventions: Device: ESWT
- Sham extracorporeal shock wave therapy (Sham Comparator): A total of 4 sessions of ESWT at 1-week intervals were applied to to the sacrococcygeal area
  Interventions: Device: ESWT

INTERVENTIONS:
Device: ESWT — Extracorporeal Shock-wave Therapy

SUMMARY:
Comparison of the efficacy of coccydynia treatment with two different probes of the ESWT device

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coccydynia by clinical examination and X-ray imaging.
* be aged ≥18 at the time of diagnosis
* be give informed consent

Exclusion Criteria:

* Malignancy
* Those who have received ESWT treatment before
* Pediatric patients
* Patients with infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 minute
  pain evaluation, higher scores mean worse outcome.
Oswestry Low Back Pain Disability Questionnaire | 5 minutes
  higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Şah, Study Director — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Yüzüncü Yıl Üniversitesi Tıp Fakültesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided